CLINICAL TRIAL: NCT04121065
Title: Interventional Not Pharmacological Study to Investigate the Role of ADA in Multiple Sclerosis PatientsTreated With an Immune-Reconstitution Therapy (2-CdA)
Brief Title: Role of ADA SNPs in Subjects With Relapsing Multiple Sclerosis (RMS)
Status: Recruiting | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, Haed of Neurology Unit, Neuromed IRCCS
Other Study IDs: ADA-MS
Record Dates: First submitted 2019-09-26; First posted 2019-10-09 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: ADA; Genetic polymorphism; Relapsing Multiple Sclerosis; Immune-reconstitution therapy; 2-CdA; single nucleotide polymorphisms; lymphopenia induced by 2-CdA treatment; ADA genetic variant rs244072; non-risk/risk allele T/C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relapsing MS patients: Single Arm: Relapsing Multiple Sclerosis patients ADA SNPs and other biomarkers analyses in blood samples.
  Interventions: Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Blood withdrawal — Blood withdrawal of maximum 60 ml performed to each enrolled patient during the study for primary and secondary endpoints evaluation.

SUMMARY:
Multiple Sclerosis (MS) is a chronic autoimmune demyelinating disease of the central nervous system (CNS), which is highly heterogeneous in terms of clinical symptoms, MS subtypes and treatment response. In each patient with MS, inflammatory, neurodegenerative and reparative processes are intermingled in different proportions, making the disease course unpredictable and the treatment approach challenging.

Although MS etiology is still unclear, many studies have demonstrated that T and B cells are crucial cellular determinants of MS pathophysiological processes. Auto-reactive T lymphocytes have been also implicated in excitotoxic synaptopathy, an early hallmark of MS recently emerged to link inflammation and neurodegeneration in a complex and inter-regulated circuit. In addition, several reports published in the last few years show the presence of a link between metabolism and immune responses. Indeed, it is now clear that cell metabolism is able to control T cell survival, growth, activation and differentiation. It has been reported that distinct metabolic pathways are able to support specific T cell activities suggesting that the delicate balance among glycolysis, fatty acid oxidation (FAO) and mitochondrial respiration drives specific effector (Tconv) and regulatory T cell (Treg) differentiation and functions.

The individual response to treatment varies widely and their use may be burdened by side effects and major adverse events. An explanation of the clinical and pharmacological individual variability can be sought in the pathological heterogeneity and in different genetic, immunological and metabolomics profiles. With this perspective, the lack of a single predictive or diagnostic test remains a great obstacle in the management of MS at most stages and in the choice of the therapy. Consequently, the availability of biomarkers that reliably capture the different aspects of the disease could be extremely useful.

DETAILED DESCRIPTION:
The therapeutic landscape for multiple sclerosis (MS) is rapidly evolving. For the past 25 years, there has been an accelerating inclusion of new immunomodulating drugs. MS immunotherapies may also be classified in a different way, into treatments that are given continuously (chronic treatments) and medications that are applied intermittently (immune reconstitution therapies [IRTs]). The principle behind the latter is depletion of the immune system that allows it to rebuild itself. An IRT by definition is given at short intermittent courses and not continuously. IRT modalities were shown to induce long-term remission of MS that, in some cases, is close to the definition of a "cure".

Most importantly, IRT using these modalities causes substantial changes in the lymphocyte repertoire after the reconstitution phase.

This is particularly true for Cladribine (2-CdA), a high efficacy therapy that selectively depletes peripheral lymphocytes, recently approved by the European Medicine Agencies for RMS patients with high activity of disease.

Lymphocytes have a high intracellular ratio of DCK to 5'-NTs compared with other cell types. Specifically, levels of DCK and the ratio of DCK to 5'-NT are high in T cells (CD4+ and CD8+), B cells, and dendritic cells but are very low in numerous non-hematologic cell types (http://biogps.gnf.org). This makes lymphocytes, mainly memory B cells, particularly sensitive to the accumulation of 2-CdA nucleotides. The intracellular accumulation of 2-CdATP leads to the incorporation of 2-CdATP into cellular DNA, disrupting the double helix structure and leading to a failure of DNA repair and synthesis. The resulting DNA strand breaks alter the cell cycle progression inducing cell death mediated by apoptosis. Although apoptosis is the most prominent mechanism of action of 2-CdA, additional mechanisms cannot be excluded. Many evidences shown that nucleotide signaling governs some of the most essential responses in immunity, ranging from antigen-driven T lymphocyte proliferation to T helper 1 (Th1) and Th2 cell differentiation, from neutrophil and macrophage chemotaxis to intracellular pathogen killing, and from NADPH-oxidase activation to IL-1β maturation and release. In addition, an analysis of lymphocytes subsets collected in the pivotal phase III trial of Cladribine showed that while T cells reduction shows some Cladribine-dose dependency, B cells have a similar reduction with both dosing schedules in the trial. Moreover, the mean number of T and B cells do not differ between patients remaining free from relapses and patients developing relapses, suggesting that efficacy of Cladribine is not strictly dependent on reduction of lymphocyte count. On the other hand, a lower lymphocyte count has been correlated with a higher risk of developing an Herpes Zoster infection, with all the events restricted and dermatomal, and most of them graded as mild or moderate. Thus, severe lymphopenia is also an important identified risk for safety. In phase III clinical trials (RCTs), 20-25% of the subjects treated with 3.5mg/kg of oral 2-CdA developed transient Grade 3-4 lymphopenia. The rate of patients who discontinued the treatment for lymphopenia was highest (12.4%) in the group that received the greatest cumulative dose of 2-CdA (CC 8.75 mg/kg) at the end of the extension phase of the CLARITY study (22). This effect has been also correlated in others disease with a reduced level of DCK mRNA and a higher level of 5'NT mRNA in lymphocytes. Though the biological activation of 2-CdA needs DCK function independently of ADA action, it cannot be excluded ADA participation in other aspects of 2-CdA mechanism of action, taking in consideration ADA crucial role in lymphocytes activation and function.

In line with this, it has been recently identified an ADA genetic variant (rs244072, non-risk/risk allele: T/C) linked to brain inflammation and MS disease severity (article in preparation), by screening more than 50 SNPs in MS-related genes of 514 MS patients and looking for association with clinical and biochemical parameters. The most striking result observed was a direct correlation between the presence of at least one risk allele and EDSS score, namely CT/CC patients show higher values of EDSS than TT patients (p=0.016).

Therefore, we hypothesize that the genetic polymorphism of ADA gene, found to correlate with MS disease severity, can also influence the 2-CdA response in term of drug sensitivity/resistance as well as side effects, like lymphocytopenia. According to the rationale, in the panorama of the current therapeutic options available to the patient MRS, Cladribine is the only immune-reconstitution therapy to have an action mechanism that interferes with that of the ADA and for this it has been selected the Cladribine as a reference treatment in clinical practice for this study.

Subjects candidate to be treated with Cladribine according to clinical practice and meeting the SmPc requirements during a pre-baseline screening period of up to -3 months before baseline (month 0), will receive an initial treatment course in week 1 and week 5 (W1-W5) as per clinical practice.

Subjects will attend visits for blood sample as per mandatory monitoring before initiating Cladribine in year 1, before initiating Cladribine in year 2, and 2 and 6 months after start of treatment in each treatment year.

The study will last 2 years for each subjects, providing five visits: screening, at month 0, at month 6, at month 12 and at month 24, according to clinical practice for MS subjects monitoring.

The primary objective of the study is to evaluate the influence of the ADA SNP rs244072 (non-risk/risk allele: T/C) on lymphopenia induced by Cladribine (2-CdA) in real world setting in patients with relapsing multiple sclerosis (RMS).

The secondary objectives are:

* To evaluate molecular, metabolic and immunological factors involved in the mode of action of Cladribine, that can influence patients' response to treatment, focusing in particular on lymphopenia;
* To collect safety and tolerability data on RMS patients treated with Cladribine;
* To assess the effect of Cladribine on progression of disability and incidence of relapses.

The study will include the collection of blood samples to investigate the primary and secondary endpoints. For these analyses, a maximum of 60 ml of blood will be collected at month 0, month 6, month 12 and month 24.

Quantitative variables will be reported as mean and standard deviation (SD) or median and Interquartile Range (Q1-Q3), Categorical variables will be reported as number (n) and percentage (%) Primary endpoints and clinical endpoints will be evaluated on all sample. Others secondary endpoint will evaluate on patients of each center unless otherwise indicated.

T Student test or Mann Whitney test will be used to compare baseline characteristics of two groups (associated with the genetic polymorphism of ADA), Chi square test o Fisher exact test when necessary, will be used for categorical variables. Shapiro Wilk test and graphics methods will be use to assess normality assumptions.

In primary endpoint analysis paired t test will be used to evaluate change in lymphocytes in each group separately. Linear mixed model will be used to compare change in two groups taking in account repetitive data for each patient (patient as random effect) group, time and group per time as fixed effects. Model assumptions will be checked, in case of they are not support logarithm data or other models will be used.

Different mixed models will be used to evaluate clinical endpoint on all sample during time.

A p value < 0.05 will be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old
2. Subjects candidate to be treated with Cladribine (2-CdA) according to clinical practice and meeting the SmPc requirements:

   * Body weight ≥ 40 Kg
   * Highly active RMS as defined by: One relapse in the previous year and at least 1 T1 Gd+ lesion or 9 or more T2 lesions, while on therapy with other disease modifying drugs (DMDs); two or more relapses in the previous year, whether on DMD treatment or not;
3. Normal lymphocyte count (absolute values 1.0-3.0×109/l) according to Cladribine local labelling;
4. EDSS score ≤5.0.

Exclusion Criteria:

1. Previous exposure to drugs such as fingolimod, natalizumab, alemtuzumab, mitoxantrone and ocrelizumab;
2. Positive hepatitis C or hepatitis B surface antigen test and/or hepatitis B core antibody test for IgG and/or IgM;
3. Current or previous history of immune deficiency disorders including a positive human immunodeficiency virus (HIV) result;
4. Currently receiving immunosuppressive or myelosuppressive therapy with, e.g., monoclonal antibodies, methotrexate, cyclophosphamide, cyclosporine or azathioprine, or chronic use of corticosteroids;
5. History of tuberculosis, presence of active tuberculosis, or latent tuberculosis;
6. Evidence or suspect of PML in MRI;
7. Active malignancy or history of malignancy.
8. Pregnant or lactating women
9. Currently receiving interferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subject with relapsing multiple sclerosis
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
1. Evaluation of lymphopenia, measured by the number of lymphocytes per cubic millimeter (mm3) and associated to ADA polymorphism | Month 0 enrollment compared to month 12; RMS patients
  Assessment of lymphopenia induced by oral Cladribine (2-CdA) treatment comparing the change in the number of pre-post treatment lymphocytes after oral Cladribine treatment at month 12 (compared with month 0), between two groups (associated with the genetic polymorphism of ADA).
  Changein the number of lymphocytes measured as number of cells per cubic millimeter (mm3), grades of lymphopenia will be assigned according to the common terminology criteria for adverse events: grade 1 (mild lymphopenia) ALC < lower limit of normal to 800/mm3, grade 2 (moderate lymphopenia) ALC < 800-500/mm3, and grade 3 (severe lymphopenia) ALC < 500-200/mm3.

SECONDARY OUTCOMES:
Genotyping of SNPs and gene expression for correlation analysis with disease effectiveness of Cladribine treatment | months 0, 6, 12 and 24
  To investigate the association between SNPs, gene expression and clinical parameters (Expanded Disability Status Score (EDSS), Kurtzke Functional System Score (KFS), 9-Hole Peg Test (9HPT), Timed 25-Foot Walk (T25FW), Symbol Digit Modality Test (SDMT), Annualized Relapses Rate (ARR) and the Percentage of "No Evidence of Disease acitivity (NEDA)) at months 0, 6, 12 and 24.
  Statistical correlations of minor allele presence of each screened SNP with gene expression and/or the clinical parameters. The significance level is established at p<0.05.
Evaluation of DCK and 5'NT genes expression | months 0, 6, 12 and 24
  Evaluation of the ratio of DCK and 5'NT genes expression at months 0, 6, 12 and 24 through the mRNA quantification by ddPCR measuring the number of copies / microliter.
Statistical correlation of EBV genotypes with responder or non-responder conditions | month 0
  Correlation of EBV genotypes with responder or non-responder conditions evaluated by clinical parameters (Expanded Disability Status Score (EDSS), Kurtzke Functional System Score (KFS), 9-Hole Peg Test (9HPT), Timed 25-Foot Walk (T25FW), Symbol Digit Modality Test (SDMT), Annualized Relapses Rate (ARR) and the Percentage of "No Evidence of Disease acitivity (NEDA)). Statistical correlations of specific EBV genotype with the clinical parameters. The significance level is established at p<0.05.
Quantification of DCK and cytosolic forms of NT5 and evaluation of CD4+ enzyme activity | months 0, 6, 12 and 24
  Assessment of cellular content of DCK and cytosolic forms of NT5 and the activity of CD4+ enzymes at months 0, 6, 12 and 24, the protein quantification will be obtained by flow cytometry measuring the relative levels of MFI (mean fluorescence intensity) values. The CD4+ enzymes will be evaluated with the luminescence-based ADP detection, measuring the ADP, based on the detection by luminometer of ATP synthesized during a luciferase/luciferin reaction and the use of an ATP-to-ADP conversion curve.
Genes expression | months 0, 6, 12 and 24
  Analysis of molecular and biochemical parameters (miRNA, mRNA and circulating exosomes), performed comparing patients responder and non-responder. miRNA and mRNA detection will be assessed by qRT-PCR, measuring the relative quantification by using the 2^(-ddCt) method.
Measure of T cell extracellular acidification rate and mitochondrial respiration | months 0, 6, 12 and 24
  Measure of T cell glycolytic (Extracellular Acidification Rate, ECAR) and mitochondrial respiration (Measurement of Oxygen Consumption Rate, OCR) at months 0, 6, 12 and 24.
Measure of metabolic profile | months 0, 6, 12 and 24
  Characterize the metabolic profile induced by Cladribine of responder/non-responder or to presence/absence of lymphopenia at months 0, 6, 12 and 24, performing a multivariate statistical analysis. The significance level is established at p<0.05.
Blood levels of B-Cell Activating Factor (BAFF) and Proliferating-Inducing Ligand | months 0, 6, 12 and 24
  Establish the blood levels of B-Cell Activating Factor (BAFF) and Proliferating-Inducing Ligand (APRIL), which have a regulatory role in B cells biology, at months 0, 6, 12 and 24.
  The proteins quantification will be measured in picograms/ milliliter.
Assessment of MFI (Mean Fluorescence Intensity) levels in NK, T and B cell subsets | months 0, 6, 12 and 24
  Assess whether Cladribine treatment affects effector and regulatory NK, T and B cell subsets at months 0, 6, 12 and 24.
  The composition of cell subpopulation will be measured by the levels of MFI.
Assessment of synaptic alterations induced by T-cell-released cytokines | month 12
  Assess a possible neuroprotective action of Cladribine in counteracting synaptic excitotoxicity by modulation of T-cell-released cytokines at month 12. The variable assessed will be the spontaneous corticostriatal excitatory currents (sEPSCs) and the spontaneous corticostriatal inhibitory currents (sEPSCs).
Assessment of disease progression measuring the change in the Expanded Disability Status Scale (EDSS)/Kurtzke | months 0, 6, 12 and 24
  Assessment of disease progression after oral Cladribine treatment by means of Expanded Disability Status Scale (EDSS)/Kurtzke at month 6, 12 and 24 compared to month 0. The variable assessed will be the change in Expanded Disability Status Scale (EDSS) compared to month 0.The EDSS is widely used in clinical trials to quantify disability and monitor the changes in the level of disability over time. The EDSS scale ranges from 0 to 10.
Assessment of Kurtzke Functional System Score (KFS) evaluating the type and severity of neurologic impairment | months 0, 6, 12 and 24
  Assessment of Functional System (KFS) at month 6, 12 and 24 compared to month 0.
  KFSS is half of a 2-part system evaluating the type and severity of neurologic impairment in MS and is based on neurologic examination of independent functions. The KFSS rates 7 functional systems (plus "other"), including pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral (or mental), and other. Each of the FSS is an ordinal clinical rating scale ranging from 0 to 5 or 6.
Assessment of upper extremity (arm and hand) function performing the 9-Hole Peg Test (9HPT) | months 0, 6, 12 and 24
  Assessment of 9-Hole Peg Test (9HPT) at month 6, 12 and 24 compared to month 0. The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and non-dominant hands are tested twice. Two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand will be executed.
Assessment of of lower extremity function, performing the Timed 25-Foot Walk test (T25FW) | months 0, 6, 12 and 24
  Assessment of Timed 25-Foot Walk (T25FW) at month 6, 12 and 24 compared to month 0.
  The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The average score of two 25-Foot Timed Walk trials will be measured.
Assessment of attention and information processing speed, performing the Symbol Digit Modality Test (SDMT) | months 0, 6, 12 and 24
  Assessment of Symbol Digit Modality Test (SDMT) at month 6, 12 and 24 compared to month 0.
  The SDMT is designed to measure divided attention and information processing speed. The examinee has 90 seconds to pair specific numbers with given geometric figures by using a reference key. The SDMT score is the sum of the correct substitutions within the 90 second interval.
Evaluation of the change in Annualized Relapse Rate (ARR). | months 0, 6, 12 and 24
  Evaluation of Annualized Relapse Rate (ARR) at month 6, 12 and 24 compared to month 0.
  Change in Annualized Relapse Rate (ARR) measured by the total number of relapses divided by the total person-time at risk of relapse.
Evaluation of Disease Activity measuring the Percentage of "No Evidence of Disease Activity" (NEDA) . | months 0, 6, 12 and 24
  Evaluation of the Percentage of "No Evidence of Disease Activity" (NEDA) at month 6, 12 and 24 compared to month 0.
  No Evidence of Disease Activity" (NEDA) will be measured as number of NEDA subjects / total number of recruited patients *100
Collection of safety and tolerability data: number of patients with treatment related adverse events classified by MedDRA | months 0, 6, 12 and 24
  Collection of safety and tolerability data on RMS patients treated with Cladribine. Number of patients with Adverse

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, Principal Investigator — IRCCS Neuromed, Pozzilli, Isernia Italy
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

REFERENCES:
- [Background] Mandolesi G, Gentile A, Musella A, Fresegna D, De Vito F, Bullitta S, Sepman H, Marfia GA, Centonze D. Synaptopathy connects inflammation and neurodegeneration in multiple sclerosis. Nat Rev Neurol. 2015 Dec;11(12):711-24. doi: 10.1038/nrneurol.2015.222. Epub 2015 Nov 20. PMID 26585978
- [Background] Procaccini C, Carbone F, Di Silvestre D, Brambilla F, De Rosa V, Galgani M, Faicchia D, Marone G, Tramontano D, Corona M, Alviggi C, Porcellini A, La Cava A, Mauri P, Matarese G. The Proteomic Landscape of Human Ex Vivo Regulatory and Conventional T Cells Reveals Specific Metabolic Requirements. Immunity. 2016 Feb 16;44(2):406-21. doi: 10.1016/j.immuni.2016.01.028. PMID 26885861
- [Background] Price AM, Dai J, Bazot Q, Patel L, Nikitin PA, Djavadian R, Winter PS, Salinas CA, Barry AP, Wood KC, Johannsen EC, Letai A, Allday MJ, Luftig MA. Epstein-Barr virus ensures B cell survival by uniquely modulating apoptosis at early and late times after infection. Elife. 2017 Apr 20;6:e22509. doi: 10.7554/eLife.22509. PMID 28425914
- [Background] Mechelli R, Manzari C, Policano C, Annese A, Picardi E, Umeton R, Fornasiero A, D'Erchia AM, Buscarinu MC, Agliardi C, Annibali V, Serafini B, Rosicarelli B, Romano S, Angelini DF, Ricigliano VA, Buttari F, Battistini L, Centonze D, Guerini FR, D'Alfonso S, Pesole G, Salvetti M, Ristori G. Epstein-Barr virus genetic variants are associated with multiple sclerosis. Neurology. 2015 Mar 31;84(13):1362-8. doi: 10.1212/WNL.0000000000001420. Epub 2015 Mar 4. PMID 25740864
- [Background] Cekic C, Linden J. Purinergic regulation of the immune system. Nat Rev Immunol. 2016 Mar;16(3):177-92. doi: 10.1038/nri.2016.4. PMID 26922909
- [Background] Samuraki M, Sakai K, Odake Y, Yoshita M, Misaki K, Nakada M, Yamada M. Multiple sclerosis showing elevation of adenosine deaminase levels in the cerebrospinal fluid. Mult Scler Relat Disord. 2017 Apr;13:44-46. doi: 10.1016/j.msard.2017.02.005. Epub 2017 Feb 6. PMID 28427701
- [Background] Dong K, Gao ZW, Zhang HZ. The role of adenosinergic pathway in human autoimmune diseases. Immunol Res. 2016 Dec;64(5-6):1133-1141. doi: 10.1007/s12026-016-8870-2. PMID 27665459
- [Background] Giovannoni G. Cladribine to Treat Relapsing Forms of Multiple Sclerosis. Neurotherapeutics. 2017 Oct;14(4):874-887. doi: 10.1007/s13311-017-0573-4. PMID 29168160
- [Background] Baker D, Herrod SS, Alvarez-Gonzalez C, Zalewski L, Albor C, Schmierer K. Both cladribine and alemtuzumab may effect MS via B-cell depletion. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 5;4(4):e360. doi: 10.1212/NXI.0000000000000360. eCollection 2017 Jul. PMID 28626781
- [Background] Ceronie B, Jacobs BM, Baker D, Dubuisson N, Mao Z, Ammoscato F, Lock H, Longhurst HJ, Giovannoni G, Schmierer K. Cladribine treatment of multiple sclerosis is associated with depletion of memory B cells. J Neurol. 2018 May;265(5):1199-1209. doi: 10.1007/s00415-018-8830-y. Epub 2018 Mar 17. PMID 29550884
- [Background] Siddiqui MK, Khurana IS, Budhia S, Hettle R, Harty G, Wong SL. Systematic literature review and network meta-analysis of cladribine tablets versus alternative disease-modifying treatments for relapsing-remitting multiple sclerosis. Curr Med Res Opin. 2018 Aug;34(8):1361-1371. doi: 10.1080/03007995.2017.1407303. Epub 2017 Nov 28. PMID 29149804
- [Background] Karussis D, Petrou P. Immune reconstitution therapy (IRT) in multiple sclerosis: the rationale. Immunol Res. 2018 Dec;66(6):642-648. doi: 10.1007/s12026-018-9032-5. PMID 30443887
- [Background] De Rosa V, Galgani M, Porcellini A, Colamatteo A, Santopaolo M, Zuchegna C, Romano A, De Simone S, Procaccini C, La Rocca C, Carrieri PB, Maniscalco GT, Salvetti M, Buscarinu MC, Franzese A, Mozzillo E, La Cava A, Matarese G. Glycolysis controls the induction of human regulatory T cells by modulating the expression of FOXP3 exon 2 splicing variants. Nat Immunol. 2015 Nov;16(11):1174-84. doi: 10.1038/ni.3269. Epub 2015 Sep 28. PMID 26414764
- [Background] Wekerle H. B cells in multiple sclerosis. Autoimmunity. 2017 Feb;50(1):57-60. doi: 10.1080/08916934.2017.1281914. PMID 28166681
- [Background] An M, Wu J, Zhu J, Lubman DM. Comparison of an Optimized Ultracentrifugation Method versus Size-Exclusion Chromatography for Isolation of Exosomes from Human Serum. J Proteome Res. 2018 Oct 5;17(10):3599-3605. doi: 10.1021/acs.jproteome.8b00479. Epub 2018 Sep 19. PMID 30192545
- [Background] Mandolesi G, De Vito F, Musella A, Gentile A, Bullitta S, Fresegna D, Sepman H, Di Sanza C, Haji N, Mori F, Buttari F, Perlas E, Ciotti MT, Hornstein E, Bozzoni I, Presutti C, Centonze D. miR-142-3p Is a Key Regulator of IL-1beta-Dependent Synaptopathy in Neuroinflammation. J Neurosci. 2017 Jan 18;37(3):546-561. doi: 10.1523/JNEUROSCI.0851-16.2016. PMID 28100738
- [Background] Parodi B, Rossi S, Morando S, Cordano C, Bragoni A, Motta C, Usai C, Wipke BT, Scannevin RH, Mancardi GL, Centonze D, Kerlero de Rosbo N, Uccelli A. Fumarates modulate microglia activation through a novel HCAR2 signaling pathway and rescue synaptic dysregulation in inflamed CNS. Acta Neuropathol. 2015 Aug;130(2):279-95. doi: 10.1007/s00401-015-1422-3. Epub 2015 Apr 29. PMID 25920452
- [Background] Gentile A, Musella A, Bullitta S, Fresegna D, De Vito F, Fantozzi R, Piras E, Gargano F, Borsellino G, Battistini L, Schubart A, Mandolesi G, Centonze D. Siponimod (BAF312) prevents synaptic neurodegeneration in experimental multiple sclerosis. J Neuroinflammation. 2016 Aug 26;13(1):207. doi: 10.1186/s12974-016-0686-4. PMID 27566665
- [Background] Harris VK, Sadiq SA. Biomarkers of therapeutic response in multiple sclerosis: current status. Mol Diagn Ther. 2014 Dec;18(6):605-17. doi: 10.1007/s40291-014-0117-0. PMID 25164543
- [Background] Comabella M, Montalban X. Body fluid biomarkers in multiple sclerosis. Lancet Neurol. 2014 Jan;13(1):113-26. doi: 10.1016/S1474-4422(13)70233-3. PMID 24331797
- [Background] Polachini CR, Spanevello RM, Casali EA, Zanini D, Pereira LB, Martins CC, Baldissareli J, Cardoso AM, Duarte MF, da Costa P, Prado AL, Schetinger MR, Morsch VM. Alterations in the cholinesterase and adenosine deaminase activities and inflammation biomarker levels in patients with multiple sclerosis. Neuroscience. 2014 Apr 25;266:266-74. doi: 10.1016/j.neuroscience.2014.01.048. Epub 2014 Feb 5. PMID 24508813